CLINICAL TRIAL: NCT07276035
Title: TMS Neuromodulation of Brain-to-Stomach Circuits in Chronic Nausea
Brief Title: Brain-Stomach Circuits in Chronic Nausea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Levinthal (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, David Levinthal, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY25100001; 1R01DK144729 (NIH)
Record Dates: First submitted 2025-11-25; First posted 2025-12-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Nausea and Vomiting Syndrome
Keywords: Chronic unexplained nausea and vomiting
MeSH Terms: conditions — Vomiting | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy subjects and CNVS subjects (Experimental): Subjects without gastric problems and subjects with Chronic Nausea and Vomiting (CNVS)
  Interventions: Device: Transcranial Magnetic Stimulation, TMS

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation, TMS — The best location for evoking an electromyographic (EMG) response of the first dorsal interosseus (FDI) muscle in left and right hand to stimulation of the primary (M1) motor cortex and the minimum stimulation intensity required to evoke a certain EMG response amplitude (Motor Threshold, MT) are determined. This serves as a reference to determine the best location and stimulation parameters to evoke GMEPs from M1 and pre-motor cortical areas.
  After identification of the GMEP hot-spot, a stomach filling task (water load test or test meal) is administered and changes in the electrogastrogram (EGG) are monitored.
  In subsequent study visits, the stomach filling task is preceded by application of neuromodulatory repetitive TMS (rTMS), targeted to the GMEP hotspot.

SUMMARY:
The goal of this study is to determine whether stimulation of the brain-stomach connection can influence stomach activity in healthy adults and in individuals suffering from chronic nausea. The main questions it aims to answer are:

* What are the best brain sites to influence the stomach?
* What are the effects of different stimulation patterns on stomach activity?
* Does the stimulation affect the sensation of nausea in participants suffering from chronic nausea?

Researchers will use a non-invasive method of brain stimulation called Transcranial Magnetic Stimulation (TMS) and will record stomach responses with skin electrodes on the abdomen.

Participants will:

* Visit the clinic at least once, and for up to 9 times more over the course of several months.
* Receive TMS while sitting in a chair similar to a dentist's chair.
* Drink water or consume a test meal during each study visit.

DETAILED DESCRIPTION:
This study will use cutaneous recordings of stomach activity (electrogastrogram, EGG) and non-invasive brain stimulation with Transcranial Magnetic Stimulation (TMS) to

1. map descending cerebral cortical-to-stomach circuitry via gastric motor-evoked potentials (GMEPs),
2. use repetitive TMS (rTMS) applied to GMEP hotspots to modulate the stomach response to a satiety task (water load or nutrient drink/meal),
3. assess differences in topography and function of cortical-to-stomach circuitry between healthy subjects and subjects suffering from chronic nausea vomiting syndrome (CNVS).

Some clinical, demographic, and autonomic data (i.e. EKG) will be recorded and used as covariates to investigate any systematic impact on the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults between ages 21-60 years old, with and without CNVS diagnosis per self-report.

Exclusion Criteria:

* body mass index (BMI) > 30
* pregnancy or intention to become pregnant
* past or present chemotherapy
* diagnosis of gastric (stomach) cancer
* any kind of gastric (stomach) surgery
* current use of GLP-1 receptor agonists (e.g. Ozempic, Trulicity)
* medications which significantly lower seizure thresholds (e.g. bupropion (Wellbutrin), fluoxetine (Prozac), or tramadol (Ultram))
* implantable devices, such as a pacemakers or nerve stimulators
* history of head injury that required hospitalization, metal in the skull, or neurologic disease such as stroke, history of seizures or history of syncope (fainting or passing out)
* neurodegenerative disease (Multiple Sclerosis, Parkinson's or Alzheimer's Disease)
* ongoing psychosis or altered cognitive status status (e.g. hearing sounds or seeing visions that are not there, or feeling confused or suffering from memory lapses)
* history of cardiovascular (i.e., heart attack), pulmonary (i.e., need for supplemental oxygen), or endocrine disease (e.g. diabetes)
* current enrollment in another study using Transcranial Magnetic Stimulation (TMS)
* current use of drugs such as amphetamines, methamphetamine, Ecstasy, Ketamine, Angel Dust/PCP, cocaine, or drinking 3 or more alcoholic drinks per day
* For healthy subjects only: chronic history of gastrointestinal symptoms (e.g., nausea, indigestion, bloating, abdominal pain)
* For CNVS subjects only: diagnosis of gastric motility disorder (e.g. gastroparesis/slow stomach emptying) or history of bowel obstruction (i.e., chronic partial small bowel obstruction)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 219 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
GMEP location | Baseline session
  Location of GMEP hotspot(s) in M1 and/or premotor areas relative to FDI hotspot
EGG power change | Each study session through study completion, up to 1 year
  Change in spectral power of the EGG in the 3 cpm frequency band associated with the gastric filling task (water load or test meal), either followed or not by neuromodulatory rTMS

SECONDARY OUTCOMES:
GMEP amplitude | Each study session through study completion, up to 1 year
  Amplitude of GMEPs at hotspot
Volume | Each study session through study completion, up to 1 year
  Volume consumed during the gastric filling task
Nausea severity (only participants suffering from chronic nausea) | Each study session through study completion, up to 1 year
  Nausea severity rating on an 11-point (0-10) Likert-scale (0=none, 10=worst possible)

CONTACTS AND LOCATIONS:
Overall Officials: David J Levinthal, MD PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Final analytic de-identified datasets will be deposited in the SPARC data repository.
Time Frame: Datasets will be deposited within 2 years of study completion for as long as the SPARC repository is active.
Access Criteria: The SPARC repository is publicly accessible.